CLINICAL TRIAL: NCT05068167
Title: Assessment of Acute Kidney Injury as a Risk Factor for Myocardial Injury After Non Cardiac Surgery in Critical Patients
Brief Title: Acute Kidney Injury as a Risk Factor for Myocardial Injury After Non Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Lecturer of Anesthesia, ICU and Pain Relief, South Egypt Cancer Institute, Assiut University, Egypt, South Egypt Cancer Institute
Other Study IDs: ACI after non cardiac surgery
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Kidney Injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury | interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Kidney function test — Creatinine twice the baseline and urine output of fewer than 0.5 ml/kg per hour for 12 hours

SUMMARY:
The incidence of acute kidney injury (AKI) postoperatively has been identified to be 21.6% in adults and 18.3% in hospitalized individuals. Surgery-related AKI is a severe complication that is related not only to short-term complications as increases in mortality rate and development of cardiac complications but also with complications on long term, such as development of chronic kidney disease. A better understanding of the mechanism of this hypthesis will lead to better management of this complication.

DETAILED DESCRIPTION:
A randomized blinded prospective study included 206patients who the candidate for major surgery at South Egypt Cancer Institute, Assiut University, Assiut, Egypt. From April 2018 till April 2019, a detailed history and careful examination, routine laboratory investigations were done, Baseline ECG was recorded 24hours before surgery and 48hours postoperative at ICU.

ELIGIBILITY:
Inclusion Criteria:

* patients who were candidates for major non cardiac surgery

Exclusion Criteria:

* chronic cardiac diseases (myocardial ischemia, heart failure), Active severe infection, pregnancy, chronic kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were candidates for major surgery in the Cancer Institute of South Egypt, Assiut University, Egypt. Patients excluded from this study were patients with chronic cardiac diseases (myocardial ischemia, heart failure, Active severe infection, pregnancy, chronic kidney disease, DM, and advanced malignancy on chemotherapy or radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Creatinine level | every 12 hours
  Creatinine twice the baseline and urine output of fewer than 0.5 ml/kg per hour for 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Alaa Ali Elzohry, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided